CLINICAL TRIAL: NCT02031731
Title: A PHASE I STUDY OF THE PHARMACOKINETICS AND SAFETY OF ONARTUZUMAB IN CHINESE PATIENTS WITH LOCALLY ADVANCED OR METASTATIC SOLID TUMORS
Brief Title: The Pharmacokinetics and Safety of Onartuzumab (MetMAb) in Chinese Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO28211
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — onartuzumab

ARMS (3):
- 4 mg/kg Onartuzumab (MetMAb) (Experimental)
  Interventions: Drug: 4 mg/kg Onartuzumab (MetMAb)
- 15 mg/kg Onartuzumab (MetMAb) (Experimental)
  Interventions: Drug: 15 mg/kg Onartuzumab (MetMAb)
- 30 mg/kg Onartuzumab (MetMAb) (Experimental)
  Interventions: Drug: 30 mg/kg Onartuzumab (MetMAb)

INTERVENTIONS:
Drug: 4 mg/kg Onartuzumab (MetMAb) — 4 mg/kg Onartuzumab (MetMAb) will be administered intravenously every 3 weeks.
  Arms: 4 mg/kg Onartuzumab (MetMAb)
Drug: 15 mg/kg Onartuzumab (MetMAb) — 15 mg/kg Onartuzumab (MetMAb) will be administered intravenously every 3 weeks.
  Arms: 15 mg/kg Onartuzumab (MetMAb)
Drug: 30 mg/kg Onartuzumab (MetMAb) — 30 mg/kg Onartuzumab (MetMAb) will be administered intravenously every 3 weeks.
  Arms: 30 mg/kg Onartuzumab (MetMAb)

SUMMARY:
This phase I study will examine the pharmacokinetics and safety of Onartuzumab (MetMAb) in chinese patients with locally advanced or metastatic solid tumors. Patients will be divided into 3 cohorts, which will each be given a different dose of MetMAb. The cohorts will be treated sequentially, starting with the lowest dose. MetMAb will be administered intravenously every 3 weeks. Patients may be treated for up to 16 cycles (21 days each) or 1 year, whichever occurs first, in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Histologically confirmed locally advanced or metastatic solid tumor that does not respond to standard treatment or for which there is no further standard treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.
* Use of effective contraception
* Life expectancy > 3 months

Exclusion Criteria:

* Brain metastasis or spinal cord compression that has not yet been definitively treated with surgery and/or radiation, and/or patients with brain metastasis that have been receiving corticosteroids.
* Previously diagnosed and treated central nervous system (CNS) metastases or spinal cord compression that has not been clinically stable for at least 2 months.
* Treatment with anti-tumor therapy within 4 weeks before the start of study treatment, with the following exception: Patients with metastatic prostate cancer on maintenance hormonal therapy, provided they meet all other eligibility criteria.
* Current, serious or uncontrolled, systemic illness.
* Recent stroke (within the past 6 months).
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs (NSAIDs).
* History of cardiovascular conditions.
* Any other disease, gastrointestinal abnormality, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
* Receipt of any investigational agent, or participation in any other clinical study, within 4 weeks before the start of study treatment.
* Major surgery within 4 weeks before the start of study treatment, without complete recovery.
* Significant traumatic injury within 3 weeks before the start of study treatment (All wounds must be fully healed prior to Day 1).
* Uncontrolled excess calcium levels.
* Known human immunodeficiency virus (HIV) infection.
* Inadequate organ function
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01-13 (Actual); Primary Completion 2014-04-14 (Actual); Study Completion 2014-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 year
Total exposure of MetMAb, as measured by area under the concentration-time curve (AUC) | Up to 1 year

SECONDARY OUTCOMES:
Incidence of anti-therapeutic antibodies against MetMAb | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Sun Yet-sen University Cancer Center, Guangzhou